CLINICAL TRIAL: NCT06153862
Title: Africa Ready Malaria Screening
Acronym: ARMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ghana (Other)
Collaborators: Shai-Osudoku District Hospital (Unknown); Kumasi Technical University (Unknown); University of Rostock (Other); University of Applied Sciences Bonn-Rhein-Sieg (Unknown); Hochschule Aalen (Unknown)
Responsible Party: Principal Investigator, Prof. Kwabena F.M. Opuni, Associate Professor, University of Ghana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GHS-ERC: 009/06/22
Record Dates: First submitted 2023-03-31; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Malaria patients (Active Comparator): Malaria patients
  Interventions: Diagnostic Test: Immuno analytical assay
- Non malaria donors (Active Comparator): Healthy individuals (donors; controls)
  Interventions: Diagnostic Test: Immuno analytical assay

INTERVENTIONS:
Diagnostic Test: Immuno analytical assay — The eluted antibodies will be used in immuno-analytical assays, such as ELISA or Western blot, or surface-coated bead-based screening platforms using either recombinantly produced MSP119 fusion protein or synthetic peptides derived from MSP119 as antigens according to standard protocols.

SUMMARY:
This study aims to develop immuno-analytical assays for testing the titres of malaria antibodies in Ghanaian patients' and/or donors' sera using a recombinantly produced MSP119 fusion protein and/or MSP119-derived synthetic peptides as antigens.

DETAILED DESCRIPTION:
In this study, immuno-analytical assays will be developed for determining the titres of malaria antibodies in sera of two groups (malaria patients and donors/healthy volunteers) using a recombinantly produced MSP119 fusion protein and/or MSP119-derived synthetic peptides as antigens. Individuals in the two groups presenting to Shai-Osudoku District hospital will be screened for signs and symptoms of malaria according to the WHO criteria. Those within the inclusion and exclusion criteria will be introduced to the study through informed consent for adults (18 years and over) or parents/guardians for children below 12 years and assent for adolescents between 12 and below 18 years, along with informed consent from their parents. Enrolled study participants' demographic data and vital signs will be captured electronically onto the CRF. Patients will have their clinical history and detailed physical examination done by the study clinicians and then be sent to the laboratory for investigations to confirm the malaria diagnosis. The results of patients will be communicated to the study clinician to commence the appropriate treatment. At the of the study, the results of all assays will be analyzed to determine if this test can be used to diagnose malaria infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed malaria (uncomplicated and complicated cases) are diagnosed by the national guidelines.
* Healthy individuals without confirmed malaria per the national guidelines.
* Adults and parents or guardians of children below 12 years willing to participate based on signed informed consent.
* Willing to give assent to adolescents between the ages of 12 and below 18 years.
* Willing to give a blood sample for the necessary investigations as explained in the informed consent.
* Willing to adhere to study procedures and a follow-up visit at the clinic, hospital, or health facility.

Exclusion Criteria:

* Anyone refusing informed consent (or assent for adolescents) to be part of the study.
* Refusal to study procedures or giving of sample for the necessary investigations.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1640 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
MSP1-19 malaria antigen | one year
  Number of participants with MSP1-19 malaria antigen as assessed by a lateral flow test kit.

SECONDARY OUTCOMES:
Anti-MSP1-19 malaria antibody | three years
  Number of participants with antiMSP1-19 malaria antibody as assessed by a lateral flow test kit.

CONTACTS AND LOCATIONS:
Overall Officials: Adjei, Study Director — Shai-Osudoku District Hospital
Locations (1):
- Shai-Osudoku District Hospital, Dodowa, Outside North America, Ghana

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in Zenodo's open data repository service (CERN). Additionally, all datasets will be stored on external drives and in-house computers. The data will be deposited as soon as possible unless there is a legitimate reason and a decision has been agreed upon to protect the data. Before the upload of datasets, a unique DOI will be assigned, which will be stated in publications to direct readers to the primary datasets. Due to the public health interest of the outcome of this work, the datasets will be shared directly with relevant stakeholders for a wider public audience. There will be restricted datasets on the subject partaking in the study to protect their identity. This restriction will not affect the dissemination of the research outputs to the broader public. Although the datasets will be stored in the Zenodo repository for long-term preservation, the in-house datasets will be stored on an external drive for additional long-term benefit.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Five years
Access Criteria: The IPD can be accessed by requesting the Principal Investigator or accessing the information directly from Zenodo's open data repository service.